CLINICAL TRIAL: NCT05312489
Title: Outcomes of Traumatic Arterial Injuries in Upper vs. Lower Extremities
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Emad Mousa Daniel, Principal Investigator, Assiut University
Other Study IDs: Vascular Trauma
Record Dates: First submitted 2022-02-16; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Vascular Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Upper extremity arterial trauma: Vascular traumatic injuries of the arterial system of the upper limbs.
- Lower extremity arterial trauma: Vascular traumatic injuries of the arterial system of the lower limbs.

SUMMARY:
The purpose of this study is to identify and compare the causes of vascular trauma at the extremities, injury characteristics, types of vascular surgical interventions, and the outcomes of traumatic vascular injuries between the upper and lower extremities.

DETAILED DESCRIPTION:
1. Primary patient assessment Patients will be clinically assessed on presentation, and resuscitation protocols will be initiated if signs of hypovolemic shock are present according to Advanced Trauma Life Support guidelines.
2. History and physical examination are the most important components of the diagnostic protocol The presence of hard signs of arterial injury

   * Absent or diminished pulses
   * Active haemorrhage
   * Large, expanding, or pulsatile hematoma
   * Bruit or thrill
   * Distal ischemia is considered an indication for surgery, and no further specific investigative measures will be taken.

   Soft signs of vascular trauma should be noted as well including
   * Small, stable hematoma
   * Unexplained hypotension
   * History of haemorrhage that is no longer present
   * Proximity of injury to major vessels
3. Investigations including:

   * The use of a hand-held Doppler examination as a diagnostic aid
   * Duplex US and CTA for imaging.
   * Lab investigations: Complete blood picture, Coagulation profile and Kidney function tests.

Options of intervention:

All vascular trauma patients will be admitted for operative management and follow up. The specific surgical intervention will be determined by the vascular surgeon according to type, site, and extent of the injury, ranging from ligation of the injured vessel to vascular graft interposition.

An injury to a peripheral artery that does not result in complete transection can be repaired depending on luminal diameter with an interrupted or continuous suturing technique. A complete transection of a peripheral artery is first managed with minimal debridement back to healthy intima at both ends then an end-to-end anastomosis or with an interposition graft of autogenous vein or prosthetics arterial graft.

ELIGIBILITY:
Inclusion Criteria:

* All peripheral arterial injuries of one or more of the extremities.

Exclusion Criteria:

* Vascular injuries limited to the venous system only.
* Vascular injuries limited to thoracic, abdominal, or neck vessels.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients fulfilling the previous criteria who are operated at Assiut University Hospital - Department of Vascular and Endovascular Surgery.
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Presence of distal pulse or signals by doppler ultrasound | Intraoperative
  Presence of distal pulse or signals by doppler ultrasound which indicates technical success of the surgery and patency of the affected artery

SECONDARY OUTCOMES:
Type of the injury in the upper extremities compared with the lower extremities | Preoperative
  blunt or penetrating injury by history and clinical examination
Presentation of the injury in the upper extremities compared with the lower extremities | Preoperative
  Bleeding or ischemia by clinical examination.
Presence of injury related complications in the upper extremities compared with the lower extremities | Preoperative
  Presence of complications(or not) like compartment syndrome, hematoma or/and associated nerve deficit by clinical examination.
Presence of postoperative complications in the upper extremities compared with the lower extremities | Postoperative for 10 days
  Presence of complications(or not) like thrombosis of the repaired vessel, pseudoaneurysm formation or/and deep vein thrombosis by clinical examination and Duplex ultrasound evaluation.
  Presence of complications(or not) like surgical site infection or/and wound dehiscence by clinical examination and culture and sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Mubarak, Study Director — Assiut University; Ashraf G Taha, Study Director — Assiut University; Osman M Ahmed, Study Director — Assiut University; Abanoub E Mousa, Principal Investigator — Assiut University

REFERENCES:
- [Background] Gallo LK, Ramos CR, Rajani RR, Benarroch-Gampel J. Management and Outcomes after Upper Versus Lower Extremity Vascular Trauma. Ann Vasc Surg. 2021 Oct;76:152-158. doi: 10.1016/j.avsg.2021.05.007. Epub 2021 Jun 18. PMID 34153492
- [Background] Feliciano DV, Moore FA, Moore EE, West MA, Davis JW, Cocanour CS, Kozar RA, McIntyre RC Jr. Evaluation and management of peripheral vascular injury. Part 1. Western Trauma Association/critical decisions in trauma. J Trauma. 2011 Jun;70(6):1551-6. doi: 10.1097/TA.0b013e31821b5bdd. No abstract available. PMID 21817992
- [Background] Feliciano DV, Moore EE, West MA, Moore FA, Davis JW, Cocanour CS, Scalea TM, McIntyre RC Jr. Western Trauma Association critical decisions in trauma: evaluation and management of peripheral vascular injury, part II. J Trauma Acute Care Surg. 2013 Sep;75(3):391-7. doi: 10.1097/TA.0b013e3182994b48. PMID 23928739
- [Background] Huber GH, Manna B. Vascular Extremity Trauma. 2023 Apr 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK536925/ PMID 30725610